CLINICAL TRIAL: NCT06874361
Title: A Prospective, Double-blind, Sham-controlled, Randomized Clinical Trial to Assess the Safety and Efficacy of the Mi-Helper Device for Acute Treatment of Migraine in an At Home Setting.
Brief Title: Cooling to Alleviate Migraine #3
Acronym: CALM3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mi-Helper, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COT-004
Record Dates: First submitted 2025-03-05; First posted 2025-03-13 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Migraine With or Without Aura; Migraine; Migraine Headache
Keywords: Neuromodulation; Device; Neuromodulation device; Decentralized
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Group I (active treatment) (Experimental): 10 liters per minute of dehumidified air administered via Mi-Helper for 15 minutes
  Interventions: Device: Mi-Helper
- Group II (sham) (Sham Comparator): 2 LPM of ambient air administered intermittently via Mi-Helper for 15 minutes
  Interventions: Device: Mi-Helper

INTERVENTIONS:
Device: Mi-Helper — The Mi-Helper device is a non-invasive, drug-free, novel therapy that uses a patented process of dry air flow across the nasal turbinates to induce a phase change (evaporation) that extracts energy (thermodynamics) causing local cooling which modulates nerves associated with pain and other symptoms of migraine. The device delivers a controlled pressure and flow of dry room temperature air along with a nebulized saline mist for added comfort and evaporative efficiency.

SUMMARY:
This is a prospective, double-blind, sham-controlled, randomized, decentralized trial. This study aims to assess the safety and efficacy of the Mi-Helper transnasal cooling device for acute treatment of migraine in an at home setting.

Adults aged 18 years to 70 years old with a diagnosis of migraine (with or without aura) for at least one year will be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 to 70 years, inclusive, of either sex at birth.
2. Lives in the contiguous United States.
3. Self-reported to be able to read and understand English sufficiently to provide electronic Informed Consent.
4. Diagnosis of migraine with or without aura for at least 1 year.
5. Individual experiences 2 to 8 migraine attacks per month documented via migraine eDiary during screening.
6. Migraine onset before 50 years of age, self-reported during screening.
7. Migraine preventive medication unchanged for 4 weeks prior to study enrollment.
8. Stated willingness to comply with all study procedures and availability for the duration of the study.
9. Individuals that own a functioning smartphone device, internet connection (Wi-Fi or data plan) and are willing to download the study app.

Exclusion Criteria:

1. Participant has difficulty distinguishing his or her migraine attacks from other types of headaches such as tension, exertion, cluster, hormonal or sinus headaches.
2. Participant has 15 or more headache days per month reported via migraine eDiary and during screening.
3. Participant using any opioid medication at the time of screening.
4. Participant has received Botox treatment, barbiturates, SPG block, nerve blocks or trigger point injections in the head or neck within the last 4 weeks of screening.
5. Participant lives at an altitude of 2000 meters or more above sea level.
6. Self-reported intolerance to intranasal therapy.
7. Self-reported recurrent epistaxis or chronic rhinosinusitis.
8. Self-reported sinus or intranasal surgery within the last 4 months of screening.
9. Self-reported history of 'complicated migraine or headaches' (i.e., hemiplegic migraine, ophthalmoplegic migraine, migrainous infarction, basilar migraine, post-traumatic headaches, post-concussion syndrome).
10. Known or suspected pregnancy as self-reported by the prospective participant at the time of screening.
11. Prospective participant unable to fully understand the consent process and provide informed consent due to either language barriers or mental capacity.
12. Self-reported diagnosis of alcohol or substance abuse disorder at the time of screening.
13. Participant with active chronic pain syndromes, such as fibromyalgia, chronic pelvic pain, or Complex Regional Pain Syndrome (CRPS); or other pain syndrome like trigeminal neuralgia.
14. Participant with severe uncontrolled psychiatric conditions or significant neurological disorders (other than migraine) that, in the Investigator's opinion, might interfere with study assessments.
15. Failure to adhere to or inability to complete Study App inputs and onboarding activities during the screening period. Participants who are not adherent during the screening period are not eligible for study entry.
16. Participation in a previous clinical study with the Mi-Helper device.
17. Participation in a migraine study or any other interventional clinical study within the3 months prior to screening.
18. Participant has an uncontrolled medical issue at the time of screening.
19. Any condition for which transnasal air flow would be contraindicated, as determined by the Principal Investigator (PI).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2025-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Ailani, MD, Principal Investigator — MedStar Georgetown Headache Center
Locations (1):
- SPRIM Pro, Indian Harbour Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the final article including results in the text, tables, figures, and appendices, will be made available after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be made available within 6 months of the study's conclusion and will remain available for at least 3 years.
Access Criteria: Researchers who provide a methodologically sound proposal to achieve results in line with the proposed outcomes will be able to obtain IPD.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group I (Active Treatment) | Group II (Sham)
Started | 77 | 79
Completed | 61 | 64
Not Completed | 16 | 15
Not completed — Physician Decision | 1 | 0
Not completed — Did not treat | 13 | 12
Not completed — Subject noncompliance | 1 | 3
Not completed — Technical issue | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (Active Treatment) | Group II (Sham) | Total
Number analyzed (Participants) | 77 | 79 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (8.6) | 40.5 (9.4) | 40.1 (9.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 11 | 12 | 23
  Female | 66 | 66 | 132
  Other or Prefer Not to Say | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 17
  Not Hispanic or Latino | 67 | 72 | 139
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 63 | 71 | 134
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 77 | 79 | 156
Highest Level of Education [Count of Participants; unit: Participants]
  Some high school | 0 | 0 | 0
  High school diploma (or GED) | 4 | 3 | 7
  Some college | 17 | 13 | 30
  Vocational school or Certificate program | 1 | 7 | 8
  College or university degree (2- or 4-year) | 34 | 23 | 57
  Graduate degree | 21 | 32 | 53
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain Freedom at 2 Hours Post Treatment
Description: Proportion of participants with a change in headache severity from mild/moderate/severe pain at baseline to no pain at 2 hours after treatment completion (if rescue medication was not used)
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Active Treatment) | Group II (Sham)
Number analyzed (Participants) | 61 | 64
Participants | 15 | 14
Statistical Analysis 1: Comparison: Group I (Active Treatment) vs Group II (Sham); Test type: Superiority; p = 0.7194, Chi-squared; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.5 to 2.7]

2. Secondary Outcome: Freedom From Most Bothersome Symptom (MBS) at 2 Hours Post Treatment
Description: Proportion of participants with a change from mild, moderate or severe symptom severity at baseline to none at 2 hours post treatment completion.
Time Frame: 2 hours
Population: The Modified Intent-to-Treat (mITT) Population included all participants who used the study intervention and completed a baseline and 2-hour post-dose pain assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Active Treatment) | Group II (Sham)
Number analyzed (Participants) | 61 | 64
Participants | 21 | 26
Statistical Analysis 1: Comparison: Group I (Active Treatment) vs Group II (Sham); Test type: Superiority; p = 0.5214, Chi-squared; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.4 to 1.7]

3. Secondary Outcome: Sustained Pain Freedom at 24 Hours Post Treatment
Description: Proportion of participants with pain freedom with no administration of rescue medication and with no recurrence of a mild/moderate/severe headache
Time Frame: 2-24 Hours
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Active Treatment) | Group II (Sham)
Number analyzed (Participants) | 61 | 64
Participants | 8 | 11
Statistical Analysis 1: Comparison: Group I (Active Treatment) vs Group II (Sham); Test type: Superiority; p = 0.5002, Chi-squared; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.3 to 2.0]

4. Secondary Outcome: Pain Relief at 2 Hours Post Treatment
Description: Proportion of participants with a change in headache severity from severe or moderate pain at baseline to mild or no pain at 2 hours post treatment completion, or from mild pain at baseline to no pain no pain at 2 hours after treatment completion (if rescue medication was not used)
Time Frame: 2 hours
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Active Treatment) | Group II (Sham)
Number analyzed (Participants) | 61 | 64
Participants | 35 | 38
Statistical Analysis 1: Comparison: Group I (Active Treatment) vs Group II (Sham); Test type: Superiority; p = 0.8202, Chi-squared; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.5 to 1.9]

5. Secondary Outcome: Participants' Global Impression of Acute Treatment Effect
Description: Measured by the Patient Global Impression of Change (PGIC), on which participants use a 7-point scale, where 1=very much improved to 7=very much worse. Scores of 1 or 2 will be considered successes.
Time Frame: 24 Hours
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Active Treatment) | Group II (Sham)
Number analyzed (Participants) | 61 | 64
Participants
  Successful Improvement | 20 | 32
  Unsuccessful Improvement | 41 | 32
Statistical Analysis 1: Comparison: Group I (Active Treatment) vs Group II (Sham); Test type: Superiority; p = 0.0471, Chi-squared; Odds Ratio, log = 0.5, 95% CI 2-sided [0.2 to 1.0]

6. Other Pre Specified Outcome: Rescue Medication Use
Description: Use of rescue medication before 2 hours post treatment completion.
Time Frame: 2 Hours
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Active Treatment) | Group II (Sham)
Number analyzed (Participants) | 61 | 64
Participants | 5 | 3

7. Other Pre Specified Outcome: Pain Freedom Immediately Post Treatment
Description: as for outcome 1
Time Frame: 0 Hours
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Active Treatment) | Group II (Sham)
Number analyzed (Participants) | 61 | 64
Participants | 6 | 5

8. Other Pre Specified Outcome: Pain Relief Immediately Post Treatment
Description: Proportion of participants with a change in headache severity from severe or moderate pain at baseline to mild or no pain at 0 hours post treatment completion, or from mild pain at baseline to no pain no pain at 0 hours after treatment completion (if rescue medication was not used)
Time Frame: 0 minutes
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Active Treatment) | Group II (Sham)
Number analyzed (Participants) | 61 | 64
Participants | 28 | 26

9. Other Pre Specified Outcome: Sustained Pain Freedom at 48 Hours Post Treatment
Description: as for outcome 3
Time Frame: 2 - 48 Hours
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Active Treatment) | Group II (Sham)
Number analyzed (Participants) | 61 | 64
Participants | 13 | 11

10. Other Pre Specified Outcome: Freedom From Most Bothersome Symptom (MBS) at Immediately Post Treatment
Description: Proportion of participants with a change from mild, moderate or severe symptom severity at baseline to none immediately post treatment completion.
Time Frame: 0 minutes
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Active Treatment) | Group II (Sham)
Number analyzed (Participants) | 61 | 64
Participants | 9 | 8

11. Other Pre Specified Outcome: Relief From Most Bothersome Symptom (MBS) Immediately Post Treatment
Description: Proportion of participants with a change from severe or moderate symptom severity at baseline to the traditional 4-point Visual Rating Scalemild or none at 0 hours, or from mild symptom severity at baseline to none at 0 hours post treatment completion (based on the traditional 4-point Visual Rating Scale)
Time Frame: 0 hours
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Active Treatment) | Group II (Sham)
Number analyzed (Participants) | 61 | 64
Participants | 28 | 31

12. Other Pre Specified Outcome: Freedom From Nausea Immediately Post Treatment
Description: Proportion of participants with a change from mild, moderate or severe symptom severity at baseline to none immediately post treatment completion (based on the traditional 4-point Visual Rating Scale)
Time Frame: 0 hours
Population: The Modified Intent-to-Treat (mITT) Population included all participants who used the study intervention and completed a baseline and 2-hour post-dose pain assessment. Only subjects who reported nausea at baseline were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Active Treatment) | Group II (Sham)
Number analyzed (Participants) | 39 | 40
Participants | 17 | 11

13. Other Pre Specified Outcome: Freedom From Photophobia Immediately Post Treatment
Description: Proportion of participants with a change from mild, moderate or severe symptom severity at baseline to none ( immediately post treatment completion.
Time Frame: 0 Hours
Population: The Modified Intent-to-Treat (mITT) Population included all participants who used the study intervention and completed a baseline and 2-hour post-dose pain assessment. Only subjects who reported photophobia at baseline were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Active Treatment) | Group II (Sham)
Number analyzed (Participants) | 51 | 60
Participants | 9 | 9

14. Other Pre Specified Outcome: Freedom From Phonophobia Immediately Post Treatment
Description: as for outcome 10
Time Frame: 0 hours
Population: The Modified Intent-to-Treat (mITT) Population included all participants who used the study intervention and completed a baseline and 2-hour post-dose pain assessment. Only subjects who reported phonophobia at baseline were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Active Treatment) | Group II (Sham)
Number analyzed (Participants) | 47 | 56
Participants | 7 | 14

15. Other Pre Specified Outcome: Freedom From Nausea at 2 Hours Post Treatment
Description: A reduction from mild, moderate or severe symptom severity at baseline to none at 2 hours post treatment completion.
Time Frame: 2 Hours
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Active Treatment) | Group II (Sham)
Number analyzed (Participants) | 39 | 40
Participants | 24 | 18

16. Other Pre Specified Outcome: Freedom From Photophobia at 2 Hours Post Treatment
Description: as for outcome 2
Time Frame: 2 Hours
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Active Treatment) | Group II (Sham)
Number analyzed (Participants) | 52 | 60
Participants | 18 | 26

17. Other Pre Specified Outcome: Freedom From Phonophobia at 2 Hours Post Treatment
Description: as for outcome 2
Time Frame: 2 Hours
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Active Treatment) | Group II (Sham)
Number analyzed (Participants) | 47 | 56
Participants | 18 | 26

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 35 day baseline period and for 48 hours post completion of treatment with the study device.
Description: Participants routinely received questionnaires via the study app at pre-set time intervals asking if they had any changes in health or adverse events. There was also an ad-hoc form available to participants throughout the study period to report any changes in health or adverse events in real time.
Arm/Group | Group I (Active Treatment) | Group II (Sham)
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/79
Other Adverse Events (participants affected / at risk) | 8/77 | 3/79
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Active Treatment) (N=77) | Group II (Sham) (N=79)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus Infection (Infections and infestations) | 1 (1) | 0 (0)
Heart Rate Increased (Investigations) | 0 (0) | 1 (1)
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-05-27): https://cdn.clinicaltrials.gov/large-docs/61/NCT06874361/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT06874361/SAP_002.pdf